CLINICAL TRIAL: NCT06353503
Title: Using Autologous Bone Marrow Aspirate Concentrate to Treat Complete Anterior Cruciate Ligament Tear.
Brief Title: Bone Marrow Aspirate Concentrate for Anterior Cruciate Ligament Tear Treatment.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: abdulmajeed hammadi (Industry)
Responsible Party: Sponsor-Investigator, abdulmajeed hammadi, GSCCBaghdad, Global Stem Cell Center, Baghdad
Organization: Global Stem Cell Center, Baghdad (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KAZ
Record Dates: First submitted 2024-03-26; First posted 2024-04-09 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Anterior Cruciate Ligament Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: single armed study open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bone marrow injection (Experimental): intra articular injection of autologous bone marrow aspirate concentrate 4cc in the injured knee under local anesthesia and ultrasound guide
  Interventions: Procedure: autologous bone marrow aspirate concentrate

INTERVENTIONS:
Procedure: autologous bone marrow aspirate concentrate — local knee joint injection of autologous bone marrow

SUMMARY:
A single armed multicenter study enrolling 20 patients using autologous bone marrow aspirate concentrate (which is done under local or general anesthesia to aspirate around 1-2 cc/kg body weight then concentration which is done by using centrifugation and special disposable kit) local injection of 4 cc per joint under ultrasonic guidance ,completely sterile field with local anesthesia.

DETAILED DESCRIPTION:
The anterior cruciate ligament (ACL) is key to the functional stability of the knee joint and is highly susceptible to injury, especially in athletes engaged in high-impact sports. Conventional treatment for partial tears may involve conservative management; however, complete tears often necessitate surgical reconstruction. In seeking alternative treatments, this study investigates the potential of bone marrow aspirate concentrate BMAC-a regenerative medicine approach-to promote healing and restore functionality to completely torn ACLs. The regenerative properties of BMAC, attributed to the presence of stem cells and growth factors, may facilitate ligament repair and regeneration. the team aim treating 1st and 2nd degree anterior cruciate ligament tear without retraction.

ELIGIBILITY:
Inclusion Criteria:

1- Confirmed diagnosis of complete or partial ACL tear via clinical examination and imaging studies.

2. Aged between 20 and 55 years, to encompass the typical age range of patients with sports-related ACL injuries.

Exclusion Criteria:

1- Patients with a history of bleeding disorders, as this could complicate the aspiration and injection procedures.

2. Individuals with a history of malignancy, due to the potential risks associated with growth factors present in BMAC.

3. Critically ill patients or those with comorbidities

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-09-27 (Estimated); Study Completion 2026-09-27 (Estimated)

PRIMARY OUTCOMES:
Functional recovery by clinical assessments of the ACL and overall knee joint stability. | every 12 weeks till 6 months
  lachman test

SECONDARY OUTCOMES:
magnetic resonance imaging of the knee joint | 6 months from starting recruitment
  to assess the degree of anterior cruciate ligament tear

CONTACTS AND LOCATIONS:
Overall Officials: abdulmajeed a hammadi, MD, Study Director — clinical stem cell studies
Locations (1):
- Ministry of Health, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No